CLINICAL TRIAL: NCT04856293
Title: A PHASE 1, OPEN-LABEL, CROSSOVER STUDY TO ESTABLISH BIOEQUIVALENCE OF AN ENCAPSULATED MICROSPHERE FORMULATION (eMS) TO THE FORMULATED CAPSULE (FC) OF CRIZOTINIB IN HEALTHY ADULT PARTICIPANTS
Brief Title: Bioequivalence Study for Crizotinib Encapsulated Microsphere Formulation (eMS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A8081074
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Healthy Participants
Keywords: Crizotinib; Encapsulated Microsphere Formulation; Healthy adult participants
MeSH Terms: interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Three Period Treatment Sequence (Experimental): Participants will receive a single 250 mg crizotinib dose of the formulated capsule(FC) formulation, a single 250 mg crizotinib dose of the encapsulated microsphere (eMS) formulation administered by sprinkling the contents into a dry glass vial, and a single 250 mg crizotinib dose of the encapsulated microsphere (eMS) formulation (administered as intact capsules)
  Interventions: Drug: Crizotinib
- Two Period Treatment Sequence (Experimental): Participants will receive a single 250 mg crizotinib dose of the formulated capsule(FC) formulation, a single 250 mg crizotinib dose of the encapsulated microsphere (eMS) formulation administered by sprinkling the contents into a dry glass vial
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Crizotinib — A single 250 mg crizotinib dose of the FC formulation
  Other Names: Treatment A
Drug: Crizotinib — A single 250 mg crizotinib dose of the encapsulated microsphere (eMS) formulation administered by sprinkling the contents into a dry glass vial
  Other Names: Treatment B
Drug: Crizotinib — A single 250 mg crizotinib dose of the single 250 mg crizotinib dose of the encapsulated microsphere (eMS) formulation (administered as intact capsules) . The intact capsules will be swallowed whole.
  Other Names: Treatment C
  Arms: Three Period Treatment Sequence

SUMMARY:
Bioequivalence study to evaluate the pharmacokinetics of a new crizotinib encapsulated microsphere (eMS) formulation

DETAILED DESCRIPTION:
In order to overcome the poor taste/palatability associated with the original oral solution formulation of crizotinib for pediatric patients, an encapsulated microsphere (eMS) formulation with improved palatability compared with the oral solution and acceptable PK characteristics was developed.

The primary objective of this study is to establish the bioequivalence of the eMS formulation to the current commercial formulation, ie, formulated capsule (FC), in adult healthy participants to support the commercialization of this new formulation.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 18 to 55 years of age, inclusive, at the time of signing the informed consent document (ICD).
2. Male and female of non-childbearing potential participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, and laboratory tests.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
4. Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
5. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in theICD and in this protocol.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease.
2. Any condition possibly affecting crizotinib absorption (eg, gastrectomy, cholecystectomy, appendectomy).
3. History of HIV infection, chronic hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb) or hepatitis C antibody (HCVAb).
4. Positive COVID-19 test.
5. History of sensitivity to heparin or heparin induced thrombocytopenia.
6. Known history of hypersensitivity to crizotinib or any components of the formulations.
7. Other medical or psychiatric condition: recent or active suicidal ideation/behavior, laboratory abnormality or conditions related to the COVID-19 pandemic that make the participant inappropriate.
8. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of crizotinib.
9. Previous administration with an investigational drug within 30 days or 5 half-lives preceding the first dose of crizotinib (whichever is longer).
10. Positive urine drug test or cotinine test.
11. Supine BP >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), BP should be repeated 2 more times.
12. Any clinically significant abnormality in 12-lead ECG, including QTcF >450 msec, Computer-interpreted ECGs may be overread by a physician experienced in reading ECGs before excluding participants.
13. AST or ALT level > (ULN); TBili level >ULN; participants with a history of Gilbert's syndrome may have direct bilirubin <= ULN; eGFR <90 ml/min/1.73 m2 per CKD-EPI equation.
14. Male participants who are unwilling or unable to comply with the contraception requirement.
15. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening.
16. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
17. Participants who currently smoke.
18. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
19. Investigator site staff members or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Plasma AUCinf after administration of the FC formulation | Day 1, Pre-dose, hour 1, 2,4,6,8,12,24,48,72,96,144 (Periods 1-3)
  Area under the plasma concentration-time profile from time zero extrapolated to infinite time
  Method of Determination:
  Linear-log trapezoidal method
Plasma Cmax after administration of the FC formulation | Day 1, Pre-dose, hour 1, 2,4,6,8,12,24,48,72,96,144 (Periods 1-3)
  Maximum plasma concentration
  Method of Determination:
  Observed directly from the data
Plasma AUClast after administration of the FC formulation | Day 1, Pre-dose, hour 1, 2,4,6,8,12,24,48,72,96,144 (Periods 1-3)
  Area under the plasma concentration time profile from time zero to the time of the last quantifiable concentration (Clast)
  Method of Determination:
  AUClast + (Clast/kel) Where Clast is the predicted plasma concentration at the last quantifiable time point and kel is the elimination rate constant estimated from the loglinear regression analysis.
Plasma AUCinf after administration of the unencapsulated eMS formulation | Day 1, Pre-dose, hour 1, 2,4,6,8,12,24,48,72,96,144 (Periods 1-3)
  Area under the plasma concentration-time profile from time zero extrapolated to infinite time
  Method of Determination:
  Linear-log trapezoidal method
Plasma Cmax after administration of the unencapsulated eMS formulation | Day 1, Pre-dose, hour 1, 2,4,6,8,12,24,48,72,96,144 (Periods 1-3)
  Maximum plasma concentration
  Method of Determination:
  Observed directly from the data
Plasma AUClast after administration of the unencapsulated eMS formulation | Day 1, Pre-dose, hour 1,2,4,6,8,12,24,48,72,96,144 (Periods 1-3)
  Area under the plasma concentration time profile from time zero to the time of the last quantifiable concentration (Clast)
  Method of Determination:
  AUClast + (Clast/kel) Where Clast is the predicted plasma concentration at the last quantifiable time point and kel is the elimination rate constant estimated from the loglinear regression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A8081074